CLINICAL TRIAL: NCT02894073
Title: Interest of a Skin Transilluminator (Such as the VeinViewer®Vision Device) for Peripheral Venous Catheter Placement in the Obese Patient: a Randomized, Controlled Pilot Study
Brief Title: Interest of a Skin Transilluminator (Such as the VeinViewer®Vision Device) for Peripheral Venous Catheter Placement in the Obese Patient
Acronym: VEINVIEW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2015_843_0010
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: General Surgery
Keywords: obese patients; peripheral venous catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): PVC placement performed in the usual manner: visual inspection of the patient's anatomy
- visualisation group (Experimental): a skin transilluminator (such as the VeinViewer®Vision) is used to guide PVC placement
  Interventions: Device: skin transilluminator

INTERVENTIONS:
Device: skin transilluminator — VeinViewer
  Arms: visualisation group

SUMMARY:
Placement of a peripheral venous catheter (PVC) is the most common invasive procedure in anaesthesia and perhaps even in the field of medicine as a whole.

DETAILED DESCRIPTION:
Placement of a peripheral venous catheter (PVC) is the most common invasive procedure in anaesthesia and perhaps even in the field of medicine as a whole. This procedure may be challenging in the obese patient - even for the most experienced healthcare professionals.

In a study, PVC placement was considered to be difficult in 46% of obese patients but only 13% of non-obese patients.

Placement of a central venous catheter is an option when PVC placement is impossible, although central access is associated with a non-negligible risk of complications (pneumothorax, infection, arterial puncture, etc.).

Facilitating peripheral venous access in obese patients should shorten the time required for PVC placement, decrease the number of perfusion attempts (a source of dissatisfaction and discomfort for the patients) and limit the use of a central venous catheter.

Although a number of novel vein visualisation devices (such as the VeinViewer®Vision from Christie Medical) have been developed to guide PVC placement, there are no literature data on the value of these devices in the management of difficult venous access in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* All obese adult patients scheduled for surgery.
* Social security coverage

Exclusion Criteria:

* Age <18.
* Contra-indication to PVC placement.
* Legal guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
duration of the PVC placement procedure | Day 0
  the time between the first puncture and the confirmation of successful PVC placement via the injection of physiological saline

CONTACTS AND LOCATIONS:
Overall Officials: Youssef ALAMI CHENTOUFI, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France